CLINICAL TRIAL: NCT07274007
Title: Management of Grade III Traumatic Splenic Injury in Hemodynamically Stable Patients ; Laparoscopic Splenectomy Versus Splenic Artery Embolization by Interventional Radiology
Brief Title: Traumatic Injury of Spleen:Laparoscopic Splenectomy Vs Splenic Artery Embolization
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ZU-IRB# 775/17-Nov-2024
Record Dates: First submitted 2025-10-01; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Grade III Traumatic Splenic Injury in Hemodynamically Stable Patients

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic Splenectomy (Active Comparator)
  Interventions: Procedure: Laparoscopic Splenectomy vs splenic Artery Embolization
- Splenic Artery Embolization (Active Comparator)
  Interventions: Procedure: Laparoscopic Splenectomy vs splenic Artery Embolization

INTERVENTIONS:
Procedure: Laparoscopic Splenectomy vs splenic Artery Embolization — Compare the quality of life and clinical outcome after using laparoscopic Splenectomy and Splenic Artery Embolization in management of grade 3 traumatic Splenic Injury in Hemodynamically Stable Patients

SUMMARY:
The goal of this clinical trial is selection of the best method in management of grade 3 traumatic Splenic Injury in Hemodynamically Stable Patients thus improving the quality of life and clinical outcome. The main questions it aims to answer are

1. Assess the quality of life and clinical outcome after using laparoscopic Splenectomy in management of grade 3 traumatic Splenic Injury in Hemodynamically Stable Patients
2. Assess the quality of life and clinical outcome after using Splenic Artery Embolization in management of grade 3 traumatic Splenic Injury in Hemodynamically Stable Patients

Researchers will compare the quality of life and clinical outcome to see if it is better using laparoscopic Splenectomy Splenic Artery Embolization

Participants will underwent laparoscopic Splenectomy or Splenic Artery Embolization and will undwent post operative follow up, follow up at outpatient clinic and will be asked about changes occurring to their daily life social activities and their quality of life

ELIGIBILITY:
Inclusion Criteria:

* Patients aged above 12 years at time of screening.
* Patients diagnosed with grade three traumatic Splenic Injury

Exclusion Criteria:

* Patients aged less than 12 years at time of screening .
* Patients diagnosed with associated visceral injury such as "liver,kidney,bowel, etc..".
* Patients diagnosed with isolated splenic injury after trauma other than grades III
* Patients contraindicated for radiological investigations or splenic artery embolization using interventional radiology such as pregnany

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with clinical complications: as pain, fever, leucocytosis, vomiting, or illeus. | 6 months
  Number of participants with clinical complications: like Pain, fever, leucocytosis, vomiting, or illeus.

SECONDARY OUTCOMES:
Recovery time: Length of postoperative hospital stay in days. | 6 months.
  Recovery time: Length of postoperative hospital stay in days.
Measuring post operative pain severity using pain severity score. | 6 months.
  Measuring post operative pain severity using pain severity score. Minimum score =1. Maximum score= 10. The lower the score the better the outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig university,Faculty of medicine, Zagazig, Egypt